CLINICAL TRIAL: NCT03461276
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, 24 Months Study in Patients With Amnestic Mild Cognitive Impairment or Very Mild Alzheimer's Disease to Investigate the Safety, Tolerability and Immune Response of Repeated Subcutaneous Injections of ABvac40
Brief Title: Safety and Immunogenicity of Repeated Doses of ABvac40 in Patients With a-MCI or Vm-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Araclon Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AB1601
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABvac40 (Experimental): Six administrations of ABvac40; the first five administered once every 4 weeks and the sixth at week 42. Each administration consists of 1mL subcutaneous injection of ABvac40.
  Interventions: Biological: ABvac40
- Placebo (Placebo Comparator): Six administrations of Placebo; the first five administered once every 4 weeks and the sixth at week 42. Each administration consists of 1mL subcutaneous injection of the vaccine's vehicle buffer without the active component.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ABvac40 — ABvac40 consists in a conjugate of Aβx-40 with a carrier protein (KLH) vehiculated in phosphate buffer containing 0.35% aluminum hydroxide as adjuvant.
  Arms: ABvac40
Biological: Placebo — Placebo consists in the vaccine's vehicle (phosphate buffer containing 0.35% aluminum hydroxide) without the conjugate.
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is the most common type of dementia, accounting for 50-75% of the estimated 47 million people with dementia worldwide. The amyloid cascade hypothesis of AD proposes that amyloid-β (Aβ) peptide accumulation in the brain, caused by an imbalance between Aβ production and clearance, is the initiating factor of a cascade ultimately leading to dementia.

Aβ peptides are generated from sequential cleavage of the amyloid precursor protein (APP), including Aβ40 and Aβ42. Aβ40 is the predominant variant (90%) among the secreted Aβ forms and although Aβ42 is more hydrophobic and prone to aggregate, and Aβ42 oligomers are regarded to be the most neurotoxic species, Aβ40 can also produce highly toxic diffusible aggregates, which can be prevented in vitro by specific anti-Aβ40 antibodies.

Several studies have proposed that a high concentration of Aβ40 in the brain distinguishes patients with AD from those who have senile plaques but are cognitively normal, pointing to the importance of Aβ40 in the onset of dementia. In keeping with this, previous studies have demonstrated that specific anti-Aβ40 antibodies label NFTs in the entorhinal cortex and the hippocampus of AD brains, and that these do not co-localize with tau NFTs, suggesting the presence of degenerating neuronal populations filled with C-terminal fragments of Aβx-40. In addition, Aβ40 is the main component of amyloid deposition around cerebral arteries causing cerebral amyloid angiopathy (CAA), which has a prevalence of about 80-90% in patients with AD (for more information see Lacosta et al. Alzheimer's Research & Therapy (2018) 10:12 DOI 10.1186/s13195-018-0340-8).

Considering those previous results suggesting that strategies targeting Aβ40 could represent novel disease-modifying therapies, we have developed ABvac40, the first active vaccine targeting the C-terminal end of the Aβ40 peptide.

The purpose of this Phase II study is to confirm in patients with a-MCI or vm-AD the level of safety and tolerability obtained in the ABvac40 Phase I clinical trial in patients with mm-AD. In addition, the study is aimed to better characterize the immune response elicited by ABvac40 and to explore its effects on AD biomarkers.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all the following inclusion criteria:

1. Male or female between 55 and 80 years of age, both inclusive, at the time of signing informed consent.
2. The patient (or legal representative, if applicable) and a close relative/caregiver must read the subject information sheet, agree to participate in the clinical trial and sign the informed consent form (the patient and a close relative/caregiver).
3. Presence of a stable caregiver to attend the patient study visits.
4. Mini-Mental Status Examination (MMSE) score between 24 and 30 points (inclusive), according to age and education level.
5. Clinical Dementia Rating (CDR) scale scoring 0.5.
6. Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Score on the Delayed Memory Index (DMI) of 85 or lower.
7. The results of the patient's MRI brain scan must be concordant with the diagnosis of clinical a-MCI or vm-AD according to the following criteria: Scheltens scale, and measurement of white matter and past haemorrhages.
8. If the patient is receiving treatment for AD, must have been stable during the two months before the selection visit.
9. Treatment for concomitant diseases must be stable during the previous month before the treatment of the study.
10. Positive assessment of the candidate by the investigator for complying with the requirements and procedures of the study.

Exclusion Criteria:

A subject meeting any of the following exclusion criteria is NOT eligible for participation in the study.

1. Known allergy to components of the vaccine or prior history of anaphylaxis, a severe allergic reaction or a history of hypersensitivity to any component of the formulation. Allergy to fish or shellfish.
2. Active infectious disease (i.e. hepatitis B, C). Positive syphilis serology.
3. History or presence of autoimmune disease, except mild eczema, rhinitis or psoriasis.
4. Presence or history of immunodeficiency (i.e. HIV).
5. Significant kidney and/or liver disease.
6. History of asthma or reactive airway disease with bronchospasm in the last 6 months, or currently on regular treatment.
7. Major uncontrolled systemic condition (e.g. diabetes, congestive heart failure, hypertension).
8. History of cancer (≤5 years since the last specific treatment). Exceptions: basocellular carcinoma.
9. Significant alterations in hematological, biochemical or urine analytical parameters, particularly those relating to levels of vitamin B12, folic acid or thyroid tests.
10. History of any other central nervous system disorder, degenerative or non-degenerative neurological or psychiatric condition that, in the investigator's opinion could be the cause of the dementia, or could explain the cognitive impairment, or that might interfere with cognitive function directly or by its treatment.
11. Geriatric Depression Scale (GDS; abbreviated version), score >5
12. Has a "yes" answer to C-SSRS suicidal ideation items 4 or 5, or any suicidal behavior within 6 months before Screening, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening.
13. History or signs of cerebrovascular disease (ischemic or haemorrhagic stroke, transient ischemic attack), or diagnosis of possible, probable or clear vascular dementia according to NINDS-AIREN criteria.
14. Presence on MRI of a relevant pattern of microvascular disease (Leukoaraiosis, Fazekas score ≥2 in the deep white matter scale or ≥4 in the global score) or more than one lacunar or territorial infarcts. Any other MRI finding that, in the opinion of the investigator, might be a relevant contributing cause of subject´s cognitive impairment. Presence of up to 3 microhemorrhages will be acceptable.
15. History of bleeding disorder or predisposing conditions, blood clotting or clinically significant abnormal results on coagulation profile at Screening, as determined by the Investigator.
16. Patients being treated with anticoagulants or antiaggregant therapy (aspirin at a prophylactic dose ≤ 325 mg daily or clopidogrel at a dose ≤75 mg daily are allowed) should not be recruited in the study.
17. Modified Hachinski Ischemic Scale, score higher than 4.
18. Surgery (with general anaesthetic) within the previous three months to be included in the trial or programed during the study period.
19. Treatment within 30 days prior to visit 0 with systemic corticosteroids or other immunosuppressant's.
20. Vaccination against influenza or any other vaccination within 2 months before first IMP dose.
21. Patients, who have previously been randomized in this trial.
22. Participation in another clinical trial within the previous 1 month to screening visit, or within the previous 12 months after the last dose to the screening visit in the case of subjects who participated in trials with a study drug whose intention was to modify the progression AD unless documentation of receipt of placebo is available. The patient cannot be included in the study if the experimental drug was an immunotherapeutic drug, including IVIG or a vaccine against Alzheimer's disease unless documentation of receipt of placebo is available.
23. Patients with alcohol or drug abuse or dependence.
24. Absolute (having a pacemaker or implantable defibrillator) or relative (bare metal stent or stent implanted in the last six months) contraindications to MRI examination. Feeling of claustrophobic do not let perform MRI or PET scan.
25. Patients unlikely to comply with the protocol (e.g., unable to return for follow-up visits).
26. Women of childbearing potential, pregnant or nursing.
27. Significant alterations in the EKG that are associated with an added risk for the patient.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- France (3):
  - Hôpital François Mitterrand, Dijon, Bourgogne-Franche-Comté
  - CHU de Montpellier, Montpellier
  - Centre de Recherche Clinique du Gérontopôle, Toulouse
- San Giovanni di Dio - Fatebenefratelli, Brescia, Italy
- Spain (18):
  - Hospital Mútua de Terrasa, Terrassa, Barcelona
  - Hospital Universitario Donosti, Donostia / San Sebastian, Guipuzcoa
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Ramón y Cajal, Colmenar Viejo, Madrid
  - CUN - Clínica Universidad de Navarra, Pamplona, Navarre
  - Cae Oroitu, Algorta, Vizcaya
  - Hospital General Universitario de Alicante, Alicante
  - Barcelona Beta Brain Research Center (BBRC), Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundació ACE, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital U. de Burgos, Burgos
  - Hospital Santa Maria de Lleida, Lleida
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lacosta AM, Pascual-Lucas M, Pesini P, Casabona D, Perez-Grijalba V, Marcos-Campos I, Sarasa L, Canudas J, Badi H, Monleon I, San-Jose I, Munuera J, Rodriguez-Gomez O, Abdelnour C, Lafuente A, Buendia M, Boada M, Tarraga L, Ruiz A, Sarasa M. Safety, tolerability and immunogenicity of an active anti-Abeta40 vaccine (ABvac40) in patients with Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase I trial. Alzheimers Res Ther. 2018 Jan 29;10(1):12. doi: 10.1186/s13195-018-0340-8. PMID 29378651
- [Derived] Pascual-Lucas M, Lacosta AM, Montanes M, Canudas J, Loscos J, Monleon I, Allue JA, Sarasa L, Fandos N, Romero J, Sarasa M, Torres M, Whyms D, Terencio J, Pinol-Ripoll G, Boada M. Safety, tolerability, immunogenicity, and efficacy of ABvac40 active immunotherapy against Abeta40 in patients with mild cognitive impairment or very mild Alzheimer's disease: A randomized, double-blind, placebo-controlled phase 2 study. Alzheimers Dement. 2025 Oct;21(10):e70776. doi: 10.1002/alz.70776. PMID 41058018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 centers in Spain (n=18), France (n=3), Italy (n=1) and Sweden (n=1) recruited subjects in this study.
  The subjects' recruitment was competitive until the required number of subjects was completed.
Pre-assignment Details: 238 subjects were screened and assessed for eligibility. 88 subjects were screening failures and an additional 16 subjects dropped out the study before being randomized. 134 subjects were randomized. Finally, 10 randomized subjects did not receive the allocated IMP. Accordingly, 124 subjects received any IMP dose, constituting the SAF analysis set.
Groups:
- Placebo Arm Part A/ABvac40 Arm Part B: Subjects received 5 monthly (every 4 weeks) immunizations with placebo plus a placebo booster shot in Part A (Placebo arm Part A). In Part B, subjects received 5 monthly (every 4 weeks) immunizations with ABvac40 plus an ABvac40 booster shot after 6 months (ABvac40 arm Part B).
- ABvac40 Arm Part A/Placebo+Booster Arm Part B: Subjects received 5 monthly (every 4 weeks) immunizations with ABvac40 plus an ABvac40 booster shot in Part A (ABvac40 arm Part A). In Part B, the subjects received placebo following this schedule, except in V13B, where they received an ABvac40 booster shot (Placebo + Booster arm Part B).
Period: Part A (18-24 Months Duration)
Arm/Group | Placebo Arm Part A/ABvac40 Arm Part B | ABvac40 Arm Part A/Placebo+Booster Arm Part B
Started | 62 | 62
Completed | 53 | 55
Not Completed | 9 | 7
Not completed — Adverse event, serious fatal | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse event, non-fatal | 3 | 1
Not completed — Patient heath status | 0 | 1
Not completed — Patient/caregiver's decision | 3 | 3
Period: Part B (18 Months Duration)
Arm/Group | Placebo Arm Part A/ABvac40 Arm Part B | ABvac40 Arm Part A/Placebo+Booster Arm Part B
Started | 37 (Out of 53 subjects completed in the Part A, 16 subjects did not continue in Part B.) | 40 (Out of 55 subjects completed in the Part A, 15 subjects did not continue in Part B.)
Completed | 33 | 38
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse event, non-fatal | 0 | 1
Not completed — Patient/caregiver's decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who received Placebo or ABvac40 during Part A.
Groups:
- Placebo Arm Part A: Subjects who received Placebo during Part A. Six administrations: the first five administered once every 4 weeks (28±3 days) and the sixth at week 42 (Visit 18), 26 weeks after the fifth. Each administration consisted of 1 mL injection of ABvac40 vehicle without its active ingredient.
- ABvac40 Arm Part A: Subjects who received ABvac40 during Part A. Six administrations: the first five administered once every 4 weeks (28±3 days) and the sixth at week 42 (Visit 18), 26 weeks after the fifth. Each administration consisted of 1 mL injection of ABvac40 (containing 0.2 mg of Aβx-40).
- Total: Total of all reporting groups
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (5.49) | 70.6 (5.95) | 70.4 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 26 | 24 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific islander | 0 | 0 | 0
  Black | 0 | 0 | 0
  Caucasian | 60 | 58 | 118
  Other | 1 | 1 | 2
  Missing | 1 | 3 | 4
Study Disease [Count of Participants; unit: Participants]
  amnestic Mild Cognitive Impairment (a-MCI) | 42 | 38 | 80
  Very Mild Alzheimer's Disease (VMAD) | 20 | 24 | 44
Amyloid-positron Emission Tomography (a-PET) Status [Count of Participants; unit: Participants]
  Positive | 45 | 47 | 92
  Negative | 17 | 15 | 32
Apolipoprotein E (ApoE) Status [Count of Participants; unit: Participants]
  Noncarriers: E2/E2 and E2/E3, E3/E3 | 24 | 24 | 48
  Carriers (Heterozygous: E2/E4, E3/E4) | 33 | 29 | 62
  Carriers (Homozygous: E4/E4) | 5 | 9 | 14
Time from Disease Diagnosis to Informed Consent [Mean (Standard Deviation); unit: months] | 14.48 (15.81) | 14.68 (13.71) | 14.58 (14.74)

OUTCOME MEASURES:

1. Primary Outcome: Average Maximal Increment of Anti-Aβ40 Antibody Signal (Optical Density [OD] in ELISA)
Description: Average maximal increment (MΔ) of plasma anti-Aβ40 antibody signal (optical density [OD] in ELISA) in each subject with regard to Baseline visit.
Time Frame: Part A (Baseline, and post-Baseline visits at Week 2A, Week 6A, Week 10A, Week 14A, Week 18A, Week 24A, Week 40A, Week 44A, Week 50A, Week 77A, and Week 104A)
Population: The Modified Intent-to-treat (mITT) analysis set comprised all subjects in the ITT analysis set who had a Baseline- and at least 1 post-Baseline anti-Aβ40 antibody assessment (optical density [OD] in ELISA without pre-adsorption).
  Analysis of the primary efficacy endpoint was carried out using the mITT analysis set. Subjects were analyzed according to their randomized treatment assignment, regardless of the treatment received.
Measure: Mean (Standard Deviation); unit: OD
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 60 | 61
OD | 0.12 (0.21) | 3.27 (0.75)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; The trial was considered successfully confirmatory regarding efficacy (immunogenicity) of ABvac40 if the average MΔ of anti-Aβ40 antibody signal (OD in ELISA) in the ABvac40 group was significantly greater than the average MΔ of anti-Aβ40 antibody signal in the Placebo group. i.e. * Null hypothesis: average MΔ anti-Aβ40 (ABvac40) ≤ average MΔ anti-Aβ40 (placebo). * Alternative hypothesis: average MΔ anti-Aβ40 (ABvac40) > average MΔ anti-Aβ40 (placebo); Test type: Superiority; p < 0.0001, t-test, 1 sided; A 1-sided t-test with a significance level of 0.025 was employed
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; Test type: Superiority — Additional test; p < 0.0001, Wilcoxon (Mann-Whitney) — 1-sided
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; The average MΔ of anti-Aβ40 antibody signal between the two treatment groups was compared using an ANCOVA model, using the MΔ anti-Aβ40 antibody signal as the dependent variable, baseline anti-Aβ40 antibody signal (OD in ELISA) as covariate and treatment group and amyloid positivity as fixed effects; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.15, 95% CI 2-sided [2.96 to 3.34], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; 1-sided t-test to compare the ABvac40 and placebo groups. The primary analysis (t-test) was repeated, using the mITT Analysis Set to test the hypothesis: * Null hypothesis: average MΔ anti-Aβ40 (ABvac40) - average MΔ anti-Aβ40 (placebo) ≤ 1.778 * Alternative hypothesis: average MΔ anti-Aβ40 (ABvac40) - average MΔ anti-Aβ40 (placebo) > 1.778 The alternative hypothesis was confirmed; Test type: Superiority; p < 0.0001, t-test, 1 sided; t-test (sensitivity hypothesis). A 1-sided t-test with a significance level of 0.025 was employed
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; The change in anti-Aβ40 antibody signal from baseline to each post-baseline efficacy visit was analyzed using a Mixed-Model Repeated Measures (MMRM), using the mITT Analysis Set. Dependent variable: change from baseline in anti-Aβ40 antibody signal. Fixed effects: treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity. Covariates: baseline anti-Aβ40 antibody signal and baseline age; Repeated measure: measures within-patient at each visit; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Subject Discontinuations Due to TEAEs
Description: Number of withdrawn subjects due to treatment-emergent adverse events (TEAEs) during the whole study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: The safety analysis set consisted of all randomized subjects who received any amount of IMP. All safety analyses used the SAF analysis set. Subjects were analyzed according to the treatment received, regardless of the treatment assigned.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Arm Part A: Subjects received 5 monthly (every 4 weeks) immunizations with placebo plus a placebo booster shot in Part A.
- ABvac40 Arm Part A: Subjects received 5 monthly (every 4 weeks) immunizations with ABvac40 plus an ABvac40 booster shot in Part A.
- ABvac40 Arm Part B: Subjects received 5 monthly (every 4 weeks) immunizations with ABvac40 plus an ABvac40 booster shot after 6 months in Part B.
- Placebo+Booster Arm Part B: Subjects received 5 monthly (every 4 weeks) immunizations with placebo plus an ABvac40 booster shot at Visit 13 in Part B.
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 4 | 2 | 0 | 1

3. Secondary Outcome: Number of Subjects With Clinically Significant Abnormalities in Physical Examination
Description: Clinically significant (CS) abnormalities in physical examination reported during the study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 4 | 1 | 4 | 2

4. Secondary Outcome: Number of Subjects With Clinically Significant Abnormalities in Neurological Examination
Description: Clinically significant (CS) abnormalities in neurological examination reported during the study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 6 | 5 | 2 | 1

5. Secondary Outcome: Number of Subjects With Clinically Significant Abnormalities in Analytical Hematology
Description: Clinically significant (CS) abnormalities in hematology parameters reported during the study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 5 | 4 | 0 | 6

6. Secondary Outcome: Number of Subjects With Clinically Significant Abnormalities in Analytical Biochemistry
Description: Clinically significant (CS) abnormalities in biochemistry parameters reported during the study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 12 | 5 | 6 | 6

7. Secondary Outcome: Number of Subjects With Clinically Significant Abnormalities in Coagulation
Description: Clinically significant (CS) abnormalities in coagulation parameters reported during the study.
Time Frame: Entire study duration (Week 0 to Week 104 in Part A, and Week 0 to Week 77 in Part B)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
Number analyzed (Participants) | 60 | 64 | 37 | 40
Participants | 4 | 1 | 3 | 2

8. Secondary Outcome: Level of Anti-Aβ40 Antibodies in CSF
Description: The change in levels of anti-Aβ40 antibodies in cerebrospinal fluid (CSF) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included the recorded outcome value as the dependent variable; treatment, protocol specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: The Intent-to-treat (ITT) analysis set consisted of all subjects randomized who received any IMP. Analysis of all secondary efficacy endpoints was carried out using the ITT analysis set. Subjects were analyzed according to their randomized treatment.
  assignment, regardless of the treatment received
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
ng/mL
  Week 50A | 0.1654 (3.86502) | 30.1826 (3.90756)
  Week 104A | 0.2014 (0.36753) | 1.2437 (0.41902)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.047, Mixed Models Analysis

9. Secondary Outcome: Level of Anti-Aβ40 Antibodies in Plasma
Description: The change in levels of anti-Aβ40 antibodies in plasma from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included the recorded outcome value as the dependent variable; treatment, protocol specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline age as covariates; and measures within-patient at each visit as a repeated measure. A compound symmetric variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 2A, Week 6A, Week 10A, Week 14A, Week 18A, Week 24A, Week 40A, Week 44A, Week 50A, Week 77A, and Week 104A)
Population: The Intent-to-treat (ITT) analysis set consisted of all subjects randomized who received any IMP. Analysis of all secondary efficacy endpoints was carried out using the ITT analysis set. Subjects were analyzed according to their randomized treatment assignment, regardless of the treatment received.
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
μg/mL
  Week 2A | 1.5580 (4.22100) | 1.5112 (4.40221)
  Week 6A | 1.5580 (4.22100) | 13.7052 (4.44801)
  Week 10A | 1.6172 (4.24276) | 44.3187 (4.41509)
  Week 14A | 1.5479 (4.24276) | 62.1946 (4.43781)
  Week 18A | 1.5789 (4.30746) | 69.8861 (4.43781)
  Week 24A | 1.5926 (4.26432) | 39.9483 (4.44151)
  Week 40A | 1.6027 (4.33264) | 14.6139 (4.48526)
  Week 44A | 1.5463 (4.35267) | 57.5771 (4.48568)
  Week 50A | 1.5993 (4.35363) | 33.5366 (4.51418)
  Week 77A | 1.5232 (4.37735) | 10.8197 (4.57100)
  Week 104A | 1.7400 (5.57743) | 10.8365 (5.82224)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.9936, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.0391, Mixed Models Analysis — MMRM - Week 6A
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 10A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p = 0.0299, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.1267, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; Test type: Other — MMRM - Week 104A; p = 0.2477, Mixed Models Analysis

10. Secondary Outcome: Level of Antibody-secreting Cells
Description: The change in levels of antibody-secreting cells from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included the recorded outcome value as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: SFU/0.5x10^6 PBMCs
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
SFU/0.5x10^6 PBMCs
  Week 2A | -0.4365 (0.37501) | 0.1868 (0.34352)
  Week 6A | -0.0906 (0.72718) | 2.3144 (0.67867)
  Week 10A | 0.3092 (0.79081) | 4.0397 (0.73611)
  Week 14A | -0.1484 (1.44968) | 7.5119 (1.36804)
  Week 18A | 0.2873 (1.02944) | 6.8827 (0.93624)
  Week 24A | 0.4827 (0.74628) | 3.6323 (0.68609)
  Week 40A | -0.5201 (0.41447) | 1.2117 (0.37194)
  Week 44A | -1.1915 (2.45820) | 10.3597 (2.23485)
  Week 50A | -0.3489 (1.07737) | 4.5496 (1.00962)
  Week 77A | -0.3969 (0.52153) | 1.8382 (0.47244)
  Week 104A | 0.1732 (0.40914) | 0.3638 (0.40349)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.2151, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.0169, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 10A; Test type: Other; p = 0.0008, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p = 0.0002, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.0023, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p = 0.0021, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p = 0.0007, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.0012, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.0018, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.738, Mixed Models Analysis

11. Secondary Outcome: Level of Aβ40 Peptides in Plasma - ABtest-IA
Description: The change in levels of anti-Aβ40 peptides in plasma (ABtest-IA) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 2A | 2.5948 (2.22120) | 3.4620 (2.16724)
  Week 6A | 3.2541 (2.66184) | 8.3468 (2.60510)
  Week 10A | 4.2669 (3.43764) | -3.3200 (3.38626)
  Week 14A | 4.7946 (4.75127) | -10.5837 (4.71154)
  Week 18A | 7.7216 (4.68637) | -13.4213 (4.61987)
  Week 24A | 6.3608 (4.06529) | -30.6595 (4.00199)
  Week 40A | 4.7336 (4.73069) | -43.2898 (4.62000)
  Week 44A | 7.4722 (5.45150) | -36.7343 (5.32882)
  Week 50A | 6.5136 (5.56714) | -36.9475 (5.43416)
  Week 77A | 9.9852 (5.15517) | -31.8000 (5.04184)
  Week 104A | 7.9352 (7.65221) | -16.5218 (7.67117)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.7623, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.1506, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 10A; Test type: Other; p = 0.1071, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p = 0.0212, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p = 0.0014, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.0251, Mixed Models Analysis

12. Secondary Outcome: Level of Aβ42 Peptides in Plasma - ABtest-IA
Description: The change in levels of anti-Aβ42 peptides in plasma (ABtest-IA) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 2A | 0.6745 (0.47690) | 0.3868 (0.47126)
  Week 6A | 1.2776 (0.77358) | 1.6248 (0.76131)
  Week 10A | 1.2091 (0.88576) | 2.1331 (0.87167)
  Week 14A | 1.6433 (0.73975) | 1.0209 (0.72987)
  Week 18A | 1.9821 (0.55465) | 1.2815 (0.54507)
  Week 24A | 2.8599 (0.72452) | 1.6125 (0.71101)
  Week 40A | 2.0361 (0.84268) | -1.2781 (0.81992)
  Week 44A | 1.7850 (1.00896) | -0.9785 (0.98520)
  Week 50A | 2.6958 (1.24460) | 0.5563 (1.21767)
  Week 77A | 2.9304 (1.15392) | 0.9045 (1.13274)
  Week 104A | 0.8402 (1.36427) | 0.5027 (1.34946)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.6515, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.7447, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 10A; Test type: Other; p = 0.4518, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p = 0.5416, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p = 0.3504, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.2109, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p = 0.0049, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p = 0.0498, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2181, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.2087, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.8599, Mixed Models Analysis

13. Secondary Outcome: Level of Aβ40 Peptides in Plasma - ABtest-MS
Description: The change in levels of anti-Aβ40 peptides in plasma (ABtest-MS) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. A compound symmetric variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 2A | 15.0554 (86.19364) | 7.2235 (87.23687)
  Week 6A | 12.9981 (86.19364) | 26.8351 (87.24290)
  Week 10A | 10.8314 (86.57079) | 123.0016 (87.42725)
  Week 14A | 10.1449 (86.57079) | 277.9974 (87.75818)
  Week 18A | 10.1987 (87.66045) | 397.6406 (88.10607)
  Week 24A | 31.0861 (86.93514) | 453.1893 (88.16061)
  Week 40A | -26.9761 (88.54373) | 377.7762 (88.44661)
  Week 44A | -28.4349 (88.50690) | 846.1633 (88.82717)
  Week 50A | -34.2153 (88.91637) | 628.9483 (88.88059)
  Week 77A | -30.9656 (89.32946) | 155.5480 (89.69327)
  Week 104A | -37.3585 (110.48329) | 85.9804 (113.05734)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.9469, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.9063, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A; MMRM - Week 10A; Test type: Other; p = 0.3418, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p = 0.0236, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p = 0.0012, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.0004, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p = 0.0008, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p < 0.0001, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.1255, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.4232, Mixed Models Analysis

14. Secondary Outcome: Level of Aβ42 Peptides in Plasma - ABtest-MS
Description: The change in levels of anti-Aβ42 peptides in plasma (ABtest-MS) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 2A | -0.1364 (1.23360) | 0.0301 (1.23242)
  Week 6A | -0.1492 (1.32406) | 1.8092 (1.32222)
  Week 10A | -1.0248 (1.33166) | 0.8740 (1.32527)
  Week 14A | 0.1680 (1.15553) | 0.4841 (1.15690)
  Week 18A | 0.6469 (1.51683) | -0.9551 (1.49962)
  Week 24A | -0.0526 (1.38574) | -1.6059 (1.38522)
  Week 40A | 2.9633 (1.71207) | 3.3472 (1.68092)
  Week 44A | 1.6060 (1.52120) | 1.9498 (1.49737)
  Week 50A | 0.2069 (1.49045) | 2.7196 (1.46044)
  Week 77A | 1.4766 (1.61328) | 4.7243 (1.58567)
  Week 104A | 4.7604 (2.18825) | 2.6870 (2.19551)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 2A; Test type: Other; p = 0.9211, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 6A; Test type: Other; p = 0.2817, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 10A; Test type: Other; p = 0.2984, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 14A; Test type: Other; p = 0.8402, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 18A; Test type: Other; p = 0.4428, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.4156, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 40A; Test type: Other; p = 0.8706, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 44A; Test type: Other; p = 0.8691, Mixed Models Analysis
Statistical Analysis 9: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2188, Mixed Models Analysis
Statistical Analysis 10: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.1448, Mixed Models Analysis
Statistical Analysis 11: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.5004, Mixed Models Analysis

15. Secondary Outcome: Cortical Fibrillary Amyloid Deposition Assessed by a-PET Scans
Description: The change in amyloid-PET (a-PET) standard centiloid global cortical area (reference Pons) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
Centiloids
  Week 50A | 1.411 (1.1203) | 3.561 (1.0918)
  Week 104A | 4.461 (1.3841) | 1.241 (1.5403)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.1058, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.0922, Mixed Models Analysis

16. Secondary Outcome: Percentage of Change in Brain Volume
Description: The percent change in brain volume from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 24A, Week 50A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
percent change
  Week 24A | -1.39 (0.157) | -1.40 (0.165)
  Week 50A | -2.05 (0.175) | -1.75 (0.187)
  Week 104A | -4.16 (0.470) | -3.11 (0.412)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.9313, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2243, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.0952, Mixed Models Analysis

17. Secondary Outcome: Percentage of Change in Hippocampal Volume
Description: The percent change in right and left hippocampal volume from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 24A, Week 50A, Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
percent change
  Week 24A - left | -1.60 (0.454) | -2.14 (0.450)
  Week 50A - left | -4.13 (0.588) | -4.24 (0.571)
  Week 104A - left | -7.13 (1.060) | -8.15 (0.965)
  Week 24A - right | -1.37 (0.442) | -1.44 (0.439)
  Week 50A - right | -3.34 (0.513) | -3.23 (0.506)
  Week 104A - right | -6.37 (1.001) | -6.49 (0.901)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A - left; Test type: Other; p = 0.3599, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A - left; Test type: Other; p = 0.8913, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A - left; Test type: Other; p = 0.4736, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A - right; Test type: Other; p = 0.9095, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A - right; Test type: Other; p = 0.8744, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A - right; Test type: Other; p = 0.9307, Mixed Models Analysis

18. Secondary Outcome: Percentage of Change in Ventricular Volume
Description: The percent change in ventricular volume from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 24A, Week 50A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
percent change
  Week 24A | 5.30 (0.584) | 5.94 (0.573)
  Week 50A | 10.63 (0.809) | 10.21 (0.819)
  Week 104A | 22.51 (1.887) | 21.26 (1.848)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.3982, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.7035, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.6334, Mixed Models Analysis

19. Secondary Outcome: Level of Aβ42 Peptides in CSF
Description: The change in levels of Aβ42 peptides in cerebrospinal fluid (CSF) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | 29.0 (19.40) | -2.0 (19.79)
  Week 104A | -15.3 (22.51) | 4.0 (25.82)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2193, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.5543, Mixed Models Analysis

20. Secondary Outcome: Level of Aβ40 Peptides in CSF
Description: The change in levels of Aβ40 peptides in cerebrospinal fluid (CSF) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | -62.3 (173.57) | -141.8 (180.07)
  Week 104A | -652.4 (227.08) | -192.5 (260.67)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.7324, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.1719, Mixed Models Analysis

21. Secondary Outcome: Aβ42/Aβ40 Ratio in CSF
Description: The change in Aβ42/Aβ40 ratio in cerebrospinal fluid (CSF) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
Ratio
  Week 50A | 0.0005 (0.00135) | 0.0009 (0.00129)
  Week 104A | 0.0016 (0.00183) | 0.0020 (0.00205)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.7977, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.8828, Mixed Models Analysis

22. Secondary Outcome: Level of Total Tau in CSF
Description: The change in levels of total Tau in cerebrospinal fluid (CSF) from baseline to each applicable postbaseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | 23.4 (12.20) | 27.6 (12.39)
  Week 104A | 25.9 (14.20) | 14.7 (16.38)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.7954, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.5895, Mixed Models Analysis

23. Secondary Outcome: Level of p-Tau 181 in CSF
Description: The change in levels of p-Tau 181 in cerebrospinal fluid (CSF) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | 2.43 (1.684) | 3.15 (1.697)
  Week 104A | 1.55 (2.387) | 0.82 (2.634)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.743, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.832, Mixed Models Analysis

24. Secondary Outcome: Level of Neurofilament Light in CSF
Description: The change in levels of neurofilament light in cerebrospinal fluid (CSF) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, treatment-by-visit interaction, and amyloid positivity as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | 59.36 (76.513) | 181.20 (78.606)
  Week 104A | 317.11 (190.948) | 276.14 (216.781)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2283, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.886, Mixed Models Analysis

25. Secondary Outcome: Level of Neurogranin in CSF
Description: The change in levels of neurogranin in cerebrospinal fluid (CSF) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The MMRM included change from baseline in the efficacy parameter as the dependent variable; treatment, protocol-specified visits, and treatment-by-visit interaction as the fixed effects; baseline efficacy parameter and baseline age as covariates; and measures within-patient at each visit as a repeated measure. An unstructured variance-covariance matrix was used. The following factors may also have be included in the model: ApoE carrier status, baseline use of AD symptomatic medication and clinical subgroup - MCI or vmAD, if found to be significantly associated with the response measure (p < 0.15).
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
pg/mL
  Week 50A | -4.69 (8.023) | -5.93 (8.328)
  Week 104A | -34.97 (13.533) | -31.13 (15.571)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.909, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.8498, Mixed Models Analysis

26. Secondary Outcome: Mini Mental State Examination Score
Description: The change in Mini Mental State Examination score (MMSE) score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  MMSE is an 11-question measure that testes five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. MMSE score ranges from 0 to 30, with lower scores indicating worst cognition.
Time Frame: Part A (baseline, and post-baseline at Week 24A, Week 50A, Week 77A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 24A | -2.15 (0.422) | -2.24 (0.420)
  Week 50A | -3.64 (0.465) | -2.65 (0.460)
  Week 77A | -4.58 (0.628) | -4.15 (0.621)
  Week 104A | -5.98 (0.816) | -4.97 (0.816)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.8711, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.1098, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.6179, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.3715, Mixed Models Analysis

27. Secondary Outcome: Clinical Dementia Rating-Sum of Boxes Score
Description: The change in clinical dementia rating-sum of boxes (CDR-SB) score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  CDR-SB is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. CDR-SB, derived as the sum of the six individual domain scores and can range from 0 to 18. The higher scores mean a worst outcome.
Time Frame: Part A (Week 24A, Week 50A, Week 77A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 24A | 0.75 (0.152) | 0.73 (0.156)
  Week 50A | 1.41 (0.222) | 1.36 (0.221)
  Week 77A | 2.12 (0.328) | 2.05 (0.325)
  Week 104A | 3.21 (0.463) | 2.90 (0.462)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.8949, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.8712, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.8748, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.6402, Mixed Models Analysis

28. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status Score
Description: The change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) total score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  RBANS assesses five cognitive domains, i.e., Immediate Memory, Visuospatial/constructional, Language, Attention, and Delayed Memory. The test consists of 12 subtests and the score on each subtest contributes to one of the five domains. Total score, which can range from 40 to 160, derived as the sum of the five domain scores. The higher scores mean a better outcome.
Time Frame: Part A (Week 24A, Week 50A, Week 77A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 24A | -1.30 (1.009) | -2.10 (1.022)
  Week 50A | -5.45 (1.076) | -5.56 (1.077)
  Week 77A | -4.71 (1.273) | -2.66 (1.255)
  Week 104A | -3.17 (1.798) | -1.33 (1.793)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.552, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.9371, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.2354, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.4608, Mixed Models Analysis

29. Secondary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living, Mild Cognitive Impairment Score
Description: The change in Alzheimer's Disease Cooperative Study - Activities of Daily Living, Mild Cognitive Impairment (ADCS-ADL MCI) total score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  ADCS-ADL MCI is a 24-item scale that includes 6 basic activities of daily living (BADL) items and 16 instrumental activities of daily living (IADL) items that provide a total score from 0-78, with a lower score indicating greater severity.
Time Frame: Part A (Week 24A, Week 50A, Week 77A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 24A | -0.99 (0.834) | -2.08 (0.844)
  Week 50A | -4.15 (1.124) | -3.78 (1.112)
  Week 77A | -6.33 (1.399) | -6.54 (1.380)
  Week 104A | -9.87 (2.002) | -10.02 (1.982)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.3246, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.8047, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A; Test type: Other; p = 0.916, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.9582, Mixed Models Analysis

30. Secondary Outcome: Trail Making Test Scores
Description: The change in Trail Making Test (TMT) scores (Trail A and Trail B) from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  TMT consists of two parts in which the patient is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the first, the targets are all numbers from 1 to 25 and the test taker needs to connect them in sequential order; in the second part, the dots go from 1 to 13 and include letters from A to L. The lower timings mean a better outcome.
Time Frame: Part A (Week 24A, Week 50A, Week 77A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
seconds
  Week 24A - Trail A | 0.54 (2.960) | -0.59 (2.939)
  Week 50A - Trail A | 11.34 (4.186) | 3.59 (4.023)
  Week 77A - Trail A | 17.42 (4.669) | 2.79 (4.425)
  Week 104A - Trail A | 20.09 (7.253) | 9.24 (6.967)
  Week 24A - Trail B | 5.43 (8.102) | -8.47 (8.464)
  Week 50A - Trail B | 18.83 (8.503) | 18.43 (9.122)
  Week 77A - Trail B | 17.13 (8.680) | 2.38 (9.762)
  Week 104A - Trail B | 20.81 (10.715) | -4.64 (11.206)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A - Trail A; Test type: Other; p = 0.777, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A - Trail A; Test type: Other; p = 0.1727, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A - Trail A; Test type: Other; p = 0.0218, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A - Trail A; Test type: Other; p = 0.2789, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A - Trail B; Test type: Other; p = 0.2261, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A - Trail B; Test type: Other; p = 0.9743, Mixed Models Analysis
Statistical Analysis 7: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 77A - Trail B; Test type: Other; p = 0.2556, Mixed Models Analysis
Statistical Analysis 8: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A - Trail B; Test type: Other; p = 0.1008, Mixed Models Analysis

31. Secondary Outcome: Investigator Global Evaluation Score
Description: The change in Investigator Global Evaluation (IGE) score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  IGE score range at baseline: 1-Good general status; 2-Slight deterioration; 3-Moderate deterioration; 4-Bad general status.
  IGE score range after baseline: 1-Marked improvement; 2-Moderate improvement; 3-Slight improvement; 4-No change; 5-Slight worsening; 6-Moderate worsening; 7-Marked worsening.
Time Frame: Part A (Week 24A, Week 50A, and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 24A | 4.02 (0.075) | 4.07 (0.077)
  Week 50A | 4.26 (0.101) | 4.21 (0.101)
  Week 104A | 4.55 (0.180) | 4.45 (0.184)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 24A; Test type: Other; p = 0.6189, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.6937, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.6981, Mixed Models Analysis

32. Secondary Outcome: Columbia Suicide Severity Rating Scale
Description: Subjects with suicidal ideation or suicidal behavior since last visit.
Time Frame: Part A (Week 24A, Week 50A, Week 77A, and Week 104A)
Population: The Intent-to-treat (ITT) analysis set consisted of all subjects randomized who received any IMP. Analysis of all secondary efficacy endpoints was carried out using the ITT analysis set. Subjects were analyzed according to their randomized treatment assignment, regardless of the treatment received.
  Number of participants entered in each row differs from the overall number of participants because data from all participants were not available at each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
Participants
  Week 24A - suicidal ideation: number analyzed (Participants) | 57 | 58
  Week 24A - suicidal ideation | 1 | 1
  Week 24A - suicidal behavior: number analyzed (Participants) | 57 | 58
  Week 24A - suicidal behavior | 0 | 0
  Week 50A - suicidal ideation: number analyzed (Participants) | 56 | 58
  Week 50A - suicidal ideation | 1 | 2
  Week 50A - suicidal behavior: number analyzed (Participants) | 56 | 58
  Week 50A - suicidal behavior | 0 | 0
  Week 77A - suicidal ideation: number analyzed (Participants) | 54 | 56
  Week 77A - suicidal ideation | 1 | 4
  Week 77A - suicidal behavior: number analyzed (Participants) | 54 | 56
  Week 77A - suicidal behavior | 0 | 0
  Week 104A - suicidal ideation: number analyzed (Participants) | 26 | 25
  Week 104A - suicidal ideation | 0 | 0
  Week 104A - suicidal behavior: number analyzed (Participants) | 26 | 25
  Week 104A - suicidal behavior | 0 | 0

33. Secondary Outcome: EuroQol 5 Dimensions 5 Levels Overall Severity Index Score
Description: The change in Euroqol 5 Dimensions 5 Levels (EQ-5D-5L) - overall severity index score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  The EQ-5D-5L descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), with each dimension measured on the following increasing scale of severity: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems.
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 50A | -0.99 (1.204) | -2.71 (1.196)
  Week 104A | -3.06 (1.740) | -0.92 (1.725)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.2863, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.3703, Mixed Models Analysis

34. Secondary Outcome: EuroQol 5 Dimensions 5 Levels - Visual Analogue Scale Score
Description: The change in Euroqol 5 Dimensions 5 levels (EQ-5D-5L) - visual analogue scale (VAS) score from baseline to each applicable post-baseline efficacy visit (Part A) was analyzed using a Mixed-Model Repeated Measures (MMRM), and the ITT analysis set.
  VAS records the patient's self-rated health on a vertical scale, ranging from 100 = 'Best imaginable health state' down to 0 = 'Worst imaginable health state'.
Time Frame: Part A (Week 50A and Week 104A)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 62 | 62
score on a scale
  Week 50A | -5.20 (2.335) | -5.07 (2.289)
  Week 104A | -5.55 (3.109) | -1.84 (3.111)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 50A; Test type: Other; p = 0.9663, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; MMRM - Week 104A; Test type: Other; p = 0.3843, Mixed Models Analysis

35. Other Pre Specified Outcome: Average Maximal Increment of Anti-Aβ40 Antibody Signal (Optical Density [OD] in ELISA) - Sensitivity
Description: Average maximal increment (MΔ) of plasma anti-Aβ40 antibody signal (optical density [OD] in ELISA) in each subject with regard to Baseline visit.
  Sensitivity analyses in the PP (Part A) analysis set.
Time Frame: as for outcome 1
Population: The Per-Protocol analysis set comprised all subjects in the ITT analysis set who received all doses of the IMP (on V1, V4, V7, V10, V13 and V18 in Part A), attended the safety visit after Booster (V20 in Part A) and had no major protocol deviations that could have affected the efficacy analyses.
Measure: Mean (Standard Deviation); unit: OD
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A
Number analyzed (Participants) | 45 | 54
OD | 0.10 (0.13) | 3.29 (0.67)
Statistical Analysis 1: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 1 sided — A 1-sided t-test with a significance level of 0.025 was employed
Statistical Analysis 2: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo Arm Part A vs ABvac40 Arm Part A; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [3.02 to 3.4], Standard Error of Mean 0.09

ADVERSE EVENTS:
Time Frame: Whole study duration (Part A+Part B; up to 42 months)
Description: AEs experienced by the subjects were collected throughout the whole study.
Arm/Group | Placebo Arm Part A | ABvac40 Arm Part A | ABvac40 Arm Part B | Placebo+Booster Arm Part B
All-Cause Mortality (participants affected / at risk) | 1/60 | 1/64 | 0/37 | 0/40
Serious Adverse Events (participants affected / at risk) | 16/60 | 17/64 | 6/37 | 2/40
Other Adverse Events (participants affected / at risk) | 53/60 | 57/64 | 30/37 | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Arm Part A (N=60) | ABvac40 Arm Part A (N=64) | ABvac40 Arm Part B (N=37) | Placebo+Booster Arm Part B (N=40)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Amyloid related imaging abnormalities (Nervous system disorders) | 9 | 8 | 1 | 0 — All Amyloid related imaging abnormalities (ARIA) events were classified as ARIA-H per study protocol and conservatively interpreted.
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Arm Part A (N=60) | ABvac40 Arm Part A (N=64) | ABvac40 Arm Part B (N=37) | Placebo+Booster Arm Part B (N=40)
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 9 | 0 | 4
Hypertension (Vascular disorders) | 6 | 3 | 0 | 0
Headache (Nervous system disorders) | 7 | 5 | 3 | 3
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 2
Injection site erythema (General disorders) | 4 | 6 | 3 | 1
Injection site reaction (General disorders) | 4 | 4 | 4 | 3
Injection site swelling (General disorders) | 1 | 5 | 2 | 1
Fatigue (General disorders) | 4 | 3 | 2 | 2
Peripheral swelling (General disorders) | 1 | 1 | 4 | 1
Inflammation (General disorders) | 0 | 3 | 1 | 2
Injection site induration (General disorders) | 1 | 3 | 1 | 3
Injection site pain (General disorders) | 1 | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 7 | 10 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 4 | 1 | 1
Irritability (Psychiatric disorders) | 1 | 3 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 11 | 5 | 4
Coronavirus infection (Infections and infestations) | 1 | 4 | 6 | 9
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 4 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Depression (Psychiatric disorders) | 3 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03461276/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03461276/SAP_001.pdf